CLINICAL TRIAL: NCT04882982
Title: Caria: Digital Intervention for Menopause Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Chorus Health (Unknown)
Responsible Party: Principal Investigator, Jennifer Duffecy, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0282
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Menopause; Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caria app (Experimental): The Caria app is publically available on the Apple app store. It is an interactive native app that provides education on menopause as well as symptom tracking/feedback features, social support as well as cognitive behavioral and relaxation techniques. Participants will be given an "unlocked" version with all content available at no charge. The app sends out occasional automated emails to users to remind of features of the app and to encourage them to return to the app. Users can opt out of reminder features.
  Interventions: Behavioral: Caria app
- Menopause education (Active Comparator): Participants will receive educational material about menopause from the North American Menopause Society, a well respected menopause organization.
  Interventions: Behavioral: Menopause Education

INTERVENTIONS:
Behavioral: Caria app — App to improve symptoms of menopause
  Arms: Caria app
Behavioral: Menopause Education — Educational materials about symptoms of menopause
  Arms: Menopause education

SUMMARY:
Menopause is the time of life when menstrual cycles cease. Women typically spend 30-40% of their lives in menopause. Individual experiences of menopause vary and although some women do not experience any significant symptoms, common symptoms include vasomotor dysfunction, vaginal dryness, mood changes, sleep disturbances, urinary incontinence, cognitive changes, somatic complaints and sexual dysfunction. Reduced quality of life can occur as a result of these symptoms. A mobile app has been developed to reduce the impact of these symptoms using a variety of behavioral change techniques including education, goal setting, motivational enhancement, social support and cognitive behavioral approaches. Participants will complete self report assessments of women's symptoms and QOL at baseline, 3 weeks and 6 weeks of app use.

ELIGIBILITY:
Inclusion Criteria:

- Women with variable menstrual cycles (menopausal transition) or those who were more than 1 year from their last menstrual period (postmenopause)

Hot flash/night sweats should be experienced as problematic (as indicated by an average score of 2 or higher on three items of the Hot Flush Rating Scale

Elevated score on at least one measure - either depression (PHQ8=10 or greater, sleep (PSQI of 5 or greater) or anxiety (GAD7=10 or greater)

Own an apple device able to run the Caria app

English speaking

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants need to be experiencing menopause or the menopausal transition.
Enrollment: 150 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Hot Flush Rating Scale | 6 weeks
  A measure of self-reported hot flashes, night sweats and/or severity of hot flashes typically using a dairy to record the frequency and severity of hot flashes using a 4-point scale: mild, moderate, severe, very severe to provide a hot flash index (sum of the number of hot flashes multiplied by severity).

SECONDARY OUTCOMES:
Women's Health Questionnaire | 6 weeks
  The Women's Health Questionnaire (WHQ) is a measure of mid-aged women's emotional and physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Duffecy, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No